CLINICAL TRIAL: NCT02953431
Title: Increased Lung Volume as Controller Therapy for Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Anne Dixon, Professor of Medicine, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-061
Record Dates: First submitted 2016-04-29; First posted 2016-11-02 (Estimated); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Asthma
Keywords: Asthma; Obesity
MeSH Terms: conditions — Asthma; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Sham CPAP (Placebo Comparator): Participants will be randomized to Sham CPAP
  Interventions: Device: CPAP
- CPAP 10 (Active Comparator): Participants will be randomized to CPAP 10
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — CPAP will be administered with a CPAP machine

SUMMARY:
This is an early phase clinical trial to test the efficacy of elevating lung volume with positive expiratory pressure (CPAP) as a controller therapy for asthma in patients with a BMI ≥ 30 kg/m2.

There will be two phases to this trial.

Phase I:

In the first phase we will determine the optimal duration of CPAP that is effective as a controller therapy in asthma. Up to 9 participants will complete this this phase.

Phase II:

The 2nd phase will be a randomized double-blinded controlled trial of Sham CPAP versus CPAP 10 (using the duration of CPAP determined in phase I) as a controller therapy for asthma, and also to determine the effect o airway reactivity in healthy people with a BMI 30 kg/m2 and above. Twenty people with asthma and twenty controls will complete this phase.

DETAILED DESCRIPTION:
The effect of 10 versus 0 cmH2O CPAP on airways responsiveness to inhaled methacholine will be studied using an adaptive "3+3" phase I/II study design.

Dose Titration Phase (phase I):

The efficacy of 8 hours of CPAP on airway responsiveness will be tested in three subjects.

Efficacy will be defined as a 25% improvement in the impedance response to methacholine in all three subjects. If this occurs in all subjects, shorter durations of CPAP will be studied (4 hours then one hour).

Conversely, if "dose escalation" is required, 3 nights, then 7 nights of CPAP will be studied.

Randomized-controlled study phase (phase II):

Participants will be randomized to CPAP 10 or Sham 0. The duration of CPAP will be determined in the dose titration phase. The effect on response to inhaled methacholine, lung function and asthma control will be determined in patients with asthma and a BMI ≥ 30 kg/m2, and also in healthy controls without asthma

ELIGIBILITY:
Inclusion Criteria for people with asthma:

1. Physician diagnosis of asthma
2. PC20 to methacholine < 16 mg/ml
3. IgE < 100 IU/ml
4. Ages 18-65 years
5. BMI >=30 kg/m2

Inclusion Criteria for controls:

1. No physician diagnosis of asthma
2. PC20 to methacholine > 16 mg/ml
3. IgE < 100 IU/ml
4. Ages 18-65 years
5. BMI >=30 kg/m2

Exclusion Criteria:

1. FEV1 < 60 % predicted
2. Other significant disease that in the opinion of the investigator would interfere with study.
3. Inability to perform required testing.
4. Smoking within last 6 months.
5. ≥ 20 pack year smoking history
6. Inability to provide informed consent
7. Pregnancy
8. Known obstructive sleep apnea/ high likelihood of obstructive sleep apnea
9. Asthma exacerbation in the prior 6 weeks
10. Stoke or heart attack in the prior 3 months
11. Known aortic aneurysm
12. Renal failure
13. A known severe heart, vascular, liver, renal, or hematological disease
14. Active allergic rhinitis
15. Recent eye surgery (within the last month)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in impedance of lung in response to methacholine measured by forced oscillation | Through study completion, an average of one week
  Average change in impedance in response to methacholine in participants assigned to Sham CPAP versus CPAP 10

SECONDARY OUTCOMES:
Change in spirometric lung function (FEV1 and FVC) | Through study completion, an average of one week
  Average change in lung function in response to methacholine in participants assigned to Sham CPAP versus CPAP 10
Change in asthma control | Through study completion, an average of one week
  Average change in asthma control in response to methacholine in participants assigned to Sham CPAP versus CPAP 10

CONTACTS AND LOCATIONS:
Overall Officials: Anne Dixon, BM BCh, Principal Investigator — University of Vermont
Locations (1):
- Vermont Lung Center, Colchester, Vermont, United States

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in the archival literature, and this will include a complete description of experimental and analytical methods used. All original data will be stored and available to interested investigators with appropriate regulatory approvals in place

REFERENCES:
- [Result] Bates JH, Dixon AE. Potential role of the airway wall in the asthma of obesity. J Appl Physiol (1985). 2015 Jan 1;118(1):36-41. doi: 10.1152/japplphysiol.00684.2014. Epub 2014 Oct 23. PMID 25342709
- [Result] Chapman DG, Irvin CG, Kaminsky DA, Forgione PM, Bates JH, Dixon AE. Influence of distinct asthma phenotypes on lung function following weight loss in the obese. Respirology. 2014 Nov;19(8):1170-7. doi: 10.1111/resp.12368. Epub 2014 Aug 19. PMID 25138203
- [Result] Al-Alwan A, Bates JH, Chapman DG, Kaminsky DA, DeSarno MJ, Irvin CG, Dixon AE. The nonallergic asthma of obesity. A matter of distal lung compliance. Am J Respir Crit Care Med. 2014 Jun 15;189(12):1494-502. doi: 10.1164/rccm.201401-0178OC. PMID 24821412